CLINICAL TRIAL: NCT02675764
Title: Sensory Stimulation to Enhance Hand Function Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO42759; P20GM109040 (NIH)
Record Dates: First submitted 2016-01-25; First posted 2016-02-05 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: hand function
MeSH Terms: conditions — Stroke | interventions — Vibration; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): The experimental group receives the wrist subthreshold vibrotactile stimulation during therapy.
  Interventions: Other: Vibration; Behavioral: therapy
- Placebo (Active Comparator): The control group will wear the vibration device with no vibration.
  * Both groups cannot feel the vibration since the vibration intensity is set below the perceptible level.
  * The vibration device is a generic, commercially-available, vibrator, not particularly used for this peripheral skin stimulation purpose.
  Interventions: Other: Placebo (for vibration); Behavioral: therapy

INTERVENTIONS:
Other: Vibration — peripheral vibration at the wrist skin at an imperceptible level
  Arms: Experimental
Other: Placebo (for vibration) — No peripheral vibration at the wrist skin
  Arms: Placebo
Behavioral: therapy — standardized hand therapy program

SUMMARY:
The objective of this pilot project is to assess the impact of the novel sensory stimulation technique the investigators have developed in enhancing outcomes of hand therapy as well as the central nervous system responsiveness in chronic stroke survivors.

DETAILED DESCRIPTION:
Stroke survivors suffer from persistent hand impairment that diminishes their functional abilities and independence, despite multiple courses of rehabilitation. Sensory stimulation can prime central excitability to increase therapy outcome. The investigators developed a new sensory stimulation technique for the hand, using imperceptible vibration applied to the wrist skin. Wearable devices with a vibrating function are low cost and can be easily adopted for rehabilitation purposes to impact a wide range of patients with sensorimotor impairment. Despite the potential for clinical benefits and easy adoption for high impact, knowledge about the long-term efficacy of this new sensory stimulation technique and its underlying mechanism is limited.

The objective of this pilot project is to assess the impact of the novel sensory stimulation technique the investigators have developed in enhancing outcomes of 2-week hand therapy as well as the central nervous system responsiveness in chronic stroke survivors. This impact will be assessed in a double-blind stratified randomized controlled trial. The hypothesis is that (a) improvement in hand function will be greater for the experimental group receiving the wrist subthreshold vibrotactile stimulation during therapy compared with the control group who will wear the device with no vibration (placebo). (b) Improvement in hand function is associated with neurophysiologic measures of central nervous system responsiveness. Clinical and neurophysiologic evaluations will be performed before, immediately after, and 2 weeks after a 2 week standardized hand therapy program with the subthreshold vibrotactile stimulation to the wrist vs. sham. The investigators preliminary studies demonstrated an acute effect of the remote subthreshold vibrotactile stimulation on immediately improved clinical sensory and motor function of the hand as well as cortical excitability in healthy young adults and chronic stroke survivors in single-session studies.

The expected outcome is the demonstration that the subthreshold vibrotactile stimulation at the wrist enhances hand function, not only immediately (preliminary studies) but also as a complement to therapy in chronic stroke survivors. This project will also provide preliminary insights regarding plasticity occurring with hand therapy augmented by the subthreshold vibrotactile stimulation. This research will have a positive impact by leading to a portable sensorimotor orthosis worn at the wrist to improve hand function for patients with sensorimotor deficits.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate impairment in upper extremity function

Exclusion Criteria:

* cognitive dysfunction
* stroke<3 months
* treatment with botulinum toxin in the affected arm within 3 months of start of study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kautz, PhD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seo NJ, Woodbury ML, Bonilha L, Ramakrishnan V, Kautz SA, Downey RJ, Dellenbach BHS, Lauer AW, Roark CM, Landers LE, Phillips SK, Vatinno AA. TheraBracelet Stimulation During Task-Practice Therapy to Improve Upper Extremity Function After Stroke: A Pilot Randomized Controlled Study. Phys Ther. 2019 Mar 1;99(3):319-328. doi: 10.1093/ptj/pzy143. PMID 30690609

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental (Therapy + Stimulation): The experimental group receives the wrist subthreshold vibrotactile stimulation during therapy.
  Vibration: peripheral vibration at the wrist skin at an imperceptible level
  therapy: standardized hand therapy program
- Placebo (Therapy + Stimulation Placebo): The control group wears the vibration device with no vibration during therapy.
  Placebo (for vibration): No peripheral vibration at the wrist skin
  therapy: standardized hand therapy program
Period: Overall Study
Arm/Group | Experimental (Therapy + Stimulation) | Placebo (Therapy + Stimulation Placebo)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The control group will wear the vibration device with no vibration.
  * Both groups cannot feel the vibration since the vibration intensity is set below the perceptible level.
  * The vibration device is a generic, commercially-available, vibrator, not particularly used for this peripheral skin stimulation purpose.
  Placebo (for vibration): No peripheral vibration at the wrist skin
  therapy: standardized hand therapy program
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10) | 64 (8) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
baseline hand motor function (Box and Block Test score) [Mean (Standard Deviation); unit: blocks] — This test measures the number of blocks that a participant moved in a minute. The scale ranges from 0 to a positive number. Higher numbers represent better outcomes.
  blocks | 29 (15) | 28 (11) | 29 (12)

OUTCOME MEASURES:

1. Primary Outcome: Box and Block Test (BBT) About a Week After the 2-week Intervention
Description: Change in hand motor function as measured by the Box and Block Test. This test measures the number of blocks that a participant moved in a minute. The scale ranges from 0 to a positive number. Higher numbers represent better outcomes.
Time Frame: post intervention (about a week after the 2-week therapy, or week 3) compared to baseline (before 2-week therapy)
Measure: Mean (Standard Error); unit: change in # of blocks
Groups:
- Placebo (Therapy + Stimulation Placebo): The control group wears the vibration device with no vibration.
  Placebo (for vibration): No peripheral vibration at the wrist skin
  therapy: standardized hand therapy program
Arm/Group | Experimental (Therapy + Stimulation) | Placebo (Therapy + Stimulation Placebo)
Number analyzed (Participants) | 6 | 6
change in # of blocks | 6 (.8) | -2 (.7)

2. Primary Outcome: Box and Block Test (BBT) at Least 2 Weeks After the 2-week Intervention
Description: as for outcome 1
Time Frame: follow up (at least 2 weeks after the 2-week therapy, or week 5) compared to baseline (before 2-week therapy)
Measure: Mean (Standard Error); unit: change in # of blocks
Arm/Group | Experimental (Therapy + Stimulation) | Placebo (Therapy + Stimulation Placebo)
Number analyzed (Participants) | 6 | 6
change in # of blocks | 4 (.8) | 0.5 (.8)

3. Primary Outcome: WMFT About a Week After the 2-week Intervention
Description: change in hand motor function as measured by the Wolf Motor Function Test hand items time. This test measures time to complete movements in seconds. More negative values represent greater reduction in time and thus better outcomes.
Time Frame: post intervention (about a week after the 2-week therapy, or week 3) compared to baseline (before 2-week therapy)
Measure: Mean (Standard Error); unit: change in ln(sec)
Arm/Group | Experimental (Therapy + Stimulation) | Placebo (Therapy + Stimulation Placebo)
Number analyzed (Participants) | 6 | 6
change in ln(sec) | -0.19 (0.07) | 0.00 (0.07)

4. Primary Outcome: WMFT at Least 2 Weeks After the 2-week Intervention
Description: as for outcome 3
Time Frame: follow up (2 weeks after the 2-week therapy, or week 5) compared to baseline (before 2-week therapy)
Measure: Mean (Standard Error); unit: change in ln(sec)
Arm/Group | Experimental (Therapy + Stimulation) | Placebo (Therapy + Stimulation Placebo)
Number analyzed (Participants) | 6 | 6
change in ln(sec) | -0.090 (0.074) | -0.089 (0.074)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 5 weeks.
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02675764/Prot_SAP_000.pdf